CLINICAL TRIAL: NCT05651984
Title: Comparative Analysis of Communication Board and Eye Tracking in Intensive Care Mechanically Ventilated Patients
Brief Title: Communication Strategies for Mechanically Ventilated Patients in Intensive Care Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: CHU de Charleroi (Other); University Hospital, Tours (Other)
Responsible Party: Principal Investigator, Emilie Szymkowicz, ICU nurse, University of Liege
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: B707201837671
Record Dates: First submitted 2022-12-02; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Mechanical Ventilation Complication; Communication, Nonverbal
Keywords: Intensive care unit; Mechanical ventilation; Alternative communication; Eye tracking; Communication board
MeSH Terms: conditions — Nonverbal Communication | interventions — Eye-Tracking Technology

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison of 2 "treatments" divided into 2 time periods, so as to constitute 4 experimental conditions. The order of the treatments allocation, organised according to 2 sequences (A-B and B-A), induces a randomisation of the included patients into 2 groups. The wash-out period between the 2 periods is not applicable in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication board (Active Comparator): The communication board consists of a printed paper interface with a size of 42 x 30 cm.
  Interventions: Device: Comparison between communication board and eye tracking
- Eye tracking (Experimental): The eye tracking device combines a laptop computer with a screen size of 29 x 16 cm, an eye tracker (PCEye Mini, Tobii dynavox, Danderyd, Sweden), an interface generated by a communication software (Communicator 5, Tobii dynavox) and a telescopic support.
  Interventions: Device: Comparison between communication board and eye tracking

INTERVENTIONS:
Device: Comparison between communication board and eye tracking — The comparison between the communication board and eye tracking, conducted as a crossover, generates a randomization of the patients (from the cross-sectional part) into two groups and the communication interfaces were divided into two time periods: group A received eye tracking/communication board sequence and group B received communication board/eye tracking sequence.

SUMMARY:
This prospective study consisted of (1) a descriptive cross-sectional part describing communication difficulties related to mechanical ventilation as experienced by intensive care professionals and patients, and (2) an experimental randomized crossover part comparing the use of a conventional low-tech communication board and a high-tech eye tracking technology-based device to improve communication effectiveness of intensive care mechanically ventilated patients.

DETAILED DESCRIPTION:
Sample size:

The health professionals sample size is estimated by convenience to 100 professionals based on the accessible population in the study site (i.e., 95% of the health professionals from the study site). The patients sample size is estimated to 44 patients based on statistical calculation (with a type 1 error rate of 5%, a type 2 error rate of 10% and an allocation ratio of 1), including two groups of 22 patients.

Intervention:

The cross-sectional part involved the healthcare professionals through the "state of the art questionnaire" and the patients through the "ease of communication scale". The crossover part then randomized the patients from the cross-sectional part into two groups and the communication interfaces were divided into two time periods: group A received eye tracking/communication board sequence and group B received communication board/eye tracking sequence. For each period, the communication interfaces were evaluated through the "intervention form". The communication board provides simple messages based on orthographic and iconic content. The eye tracking computer-based system enables the production and construction of simple or complex messages (including word processing with spelling suggestions and voice synthesis), also based on orthographic and iconic content.

Statistical analysis:

The numerical data will be analyzed quantitatively using R software (version 2016 3.5.3). The Gaussian distribution will be estimated by mean/median comparison, histogram symmetry, quantile-quantile distribution and shapiro-wilk test. Statistical analysis of the crossover variables (treatment-period interaction, period effect, and treatment effect) will be performed using the Mann-Whitney (ordinal variables) and chi-square (binary variables) nonparametric tests. A p-value less than 0.05 was considered significant. The non-numerical data will be analyzed qualitatively by thematization and categorization.

Ethics approval and consent to participate:

The study protocol was approved by the Ethics Committee of the Hospital of Liège as Central Committee and the Hospital of Charleroi as Local Committee (number: B70720183767, reference: 2018/268). The information and consent documents intended for healthcare professionals and patients were validated by both Ethics Committees. Written informed consent was obtained from all participants (healthcare professionals and patient's legal representative) included in this study. All procedures performed through this study were in accordance with the 1964 Helsinki Declaration and its later amendments.

ELIGIBILITY:
Inclusion Criteria - healthcare professionals:

* Working in the intensive care unit (study site).

Exclusion Criteria - healthcare professionals:

* Lack of consent.

Inclusion Criteria - patients:

* Being hospitalized in the intensive care unit (study site),
* Awake with a Richmond Agitation-Sedation Scale (RASS) between "restless" (+1) and "drowsy" (-1),
* Age of 18 years or older,
* French speaker.

Exclusion Criteria - patients:

* Lack of consent,
* Severe visual impairment (e.g., blindness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-02-09 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
State of the art questionnaire - communication difficulties related to mechanical ventilation as experienced by healthcare professionals. | Before the use of communication interfaces.
  Self-administered questionnaire assessing the difficulties to communicate with intubated or tracheostomized patients, the avoidance of interactions with patients, the perception of the help that could be provided by alternative communication systems and the interest in learning to use these systems.
Ease of communication scale (ECS) - communication difficulties related to mechanical ventilation as experienced by patients. | Before the use of communication interfaces.
  Multidimensional scale completed through an assisted interview and covering the difficulty to be understood; to communicate physical needs, thoughts, and feelings with notably relatives, nurses and physicians; and to ask questions about care and health status.
Quantity of messages transmitted through the communication board. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Quantity of messages transmitted through the eye tracking. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Success rate for the communication board. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Success rate for the eye tracking. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Level of satisfaction for the communication board. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Level of satisfaction for the eye tracking. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Communication content for the communication board. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Communication content for the eye tracking. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Difficulties of use related to the communcation board. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.
Difficulties of use related to the eye tracking. | During the use of communication interfaces.
  Communication effectiveness indicator, collected through the intervention form.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Ehrmann, MD, PhD, Study Director — University hospital and University of Tours; Laetitia Bodet-Contentin, MD, PhD, Study Director — University hospital and University of Tours; Yoann Marechal, MD, PhD, Principal Investigator — University hospital of Charleroi; Emilie Szymkowicz, MSc, Principal Investigator — University of Liege
Locations (1):
- University of Liège, Liège, Belgium

REFERENCES:
- [Background] Ten Hoorn S, Elbers PW, Girbes AR, Tuinman PR. Communicating with conscious and mechanically ventilated critically ill patients: a systematic review. Crit Care. 2016 Oct 19;20(1):333. doi: 10.1186/s13054-016-1483-2. PMID 27756433
- [Background] Garry J, Casey K, Cole TK, Regensburg A, McElroy C, Schneider E, Efron D, Chi A. A pilot study of eye-tracking devices in intensive care. Surgery. 2016 Mar;159(3):938-44. doi: 10.1016/j.surg.2015.08.012. Epub 2015 Sep 8. PMID 26361099
- [Background] Bodet-Contentin L, Gadrez P, Ehrmann S. Eye-tracking and speech-generating technology to improve communication with intubated intensive care unit patients: initial experience. Intensive Care Med. 2018 May;44(5):676-677. doi: 10.1007/s00134-018-5093-0. Epub 2018 Mar 3. No abstract available. PMID 29502253
- [Background] Miglietta MA, Bochicchio G, Scalea TM. Computer-assisted communication for critically ill patients: a pilot study. J Trauma. 2004 Sep;57(3):488-93. doi: 10.1097/01.ta.0000141025.67192.d9. PMID 15454792
- [Background] Maringelli F, Brienza N, Scorrano F, Grasso F, Gregoretti C. Gaze-controlled, computer-assisted communication in Intensive Care Unit: "speaking through the eyes". Minerva Anestesiol. 2013 Feb;79(2):165-75. Epub 2012 Nov 22. PMID 23174919